CLINICAL TRIAL: NCT02450331
Title: A Phase III, Open-Label, Multicenter, Randomized Study of Atezolizumab (Anti-PD-L1 Antibody) Versus Observation as Adjuvant Therapy in Patients With High-Risk Muscle-Invasive Urothelial Carcinoma After Surgical Resection
Brief Title: A Study of Atezolizumab Versus Observation as Adjuvant Therapy in Participants With High-Risk Muscle-Invasive Urothelial Carcinoma (UC) After Surgical Resection
Acronym: IMvigor010
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decided to terminate the study early because the study did not meet its primary endpoint and because the study had met its goals of providing safety and additional exploratory efficacy information for atezolizumab monotherapy in MIBC.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WO29636; 2014-005603-25 (EudraCT Number)
Record Dates: First submitted 2015-05-19; First posted 2015-05-21 (Estimated); Results first posted 2020-11-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-05

CONDITIONS: Carcinoma, Transitional Cell
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — atezolizumab

ARMS (2):
- Atezolizumab (Experimental): Participants will receive intravenous (IV) atezolizumab on Day 1 of each 21-day cycle for 16 cycles (up to 1 year).
  Interventions: Drug: Atezolizumab
- Observation (No Intervention): Participants will undergo observation starting on Day 1 for 16 cycles (up to 1 year).

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered at a dose of 1200 milligrams (mg).
  Other Names: TECENTRIQ®; MPDL3280A
  Arms: Atezolizumab

SUMMARY:
This Phase III, open-label, randomized, multicenter study is to evaluate the efficacy and safety of adjuvant treatment with atezolizumab compared with observation in participants with muscle-invasive UC who are at high risk for recurrence following resection. Eligible participants were randomized by a 1:1 ratio into atezolizumab group or control group.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed muscle-invasive UC (also termed transitional cell carcinoma) of the bladder or upper urinary tract (i.e., renal pelvis or ureters)
* For participants treated with prior neoadjuvant chemotherapy: tumor stage of ypT2-4a or ypN+ (ypT2-4 or ypN+ for participants with upper urinary tract UC) and M0
* For participants who have not received prior neoadjuvant chemotherapy: tumor stage of pT3-4a or pN+ (pT3-4 or pN+ for participants with upper urinary tract UC) and M0
* Representative formalin-fixed paraffin-embedded tumor specimens from surgical resection (i.e., radical cystectomy, nephroureterectomy, or lymph node dissection) in paraffin blocks (blocks preferred) or at least 15 unstained slides, with an associated pathology report, for central testing and determined to be evaluable for tumor programmed death-ligand 1 (PD-L1) expression prior to study enrollment
* Absence of residual disease and absence of metastasis, as confirmed by a negative baseline computed tomography (CT) or magnetic resonance imaging scan of the pelvis, abdomen, and chest no more than 4 weeks prior to randomization
* Full recovery from cystectomy or nephroureterectomy within 14 weeks following surgery
* Eastern Cooperative Oncology Group performance status of less than or equal to (</=) 2
* Life expectancy greater than or equal to (>/=) 12 weeks
* Adequate hematologic and end-organ function
* For women who are not postmenopausal or surgically sterile: agreement to remain abstinent or use contraceptive methods that result in a failure rate of less than (<) 1 percent (%) per year during the treatment period and for at least 5 months after the last dose of atezolizumab

Exclusion Criteria:

* Any approved anti-cancer therapy within 3 weeks prior to initiation of study treatment
* Adjuvant chemotherapy or radiation therapy for UC following surgical resection
* Treatment with any other investigational agent or participation in another clinical trial with therapeutic intent within 28 days or five half-lives of the drug prior to enrollment
* Malignancies other than UC within 5 years prior to Cycle 1, Day 1
* Pregnancy or breastfeeding
* Significant cardiovascular disease
* Severe infections within 4 weeks prior to Cycle 1, Day 1
* Major surgical procedure other than for diagnosis within 28 days prior to Cycle 1, Day 1
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the atezolizumab formulation
* History of autoimmune disease
* Prior allogeneic stem cell or solid organ transplant
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan
* Positive test for human immunodeficiency virus and/or active hepatitis B or hepatitis C or tuberculosis
* Administration of a live, attenuated vaccine within 4 weeks before Cycle 1 Day 1
* Prior treatment with cluster of differentiation 137 (CD137) agonists or immune checkpoint blockade therapies, including anti-CD40, anti-cytotoxic T-lymphocyte-associated protein 4 (anti-CTLA-4), anti-programmed death-1 (anti-PD-1), and anti-PD-L1 therapeutic antibodies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 809 (Actual)
Dates: Start 2015-10-05 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2022-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (186):
- United States (41):
  - HonorHealth Research Institute - Pima - Virginia G. Piper Cancer Care Network, Scottsdale, Arizona
  - UCLA, Los Angeles, California
  - USC Norris Cancer Center, Los Angeles, California
  - Stanford University Medical Center, Palo Alto, California
  - University Of Colorado, Aurora, Colorado
  - The Urology Center of Colorado, Denver, Colorado
  - Yale Cancer Center; Medical Oncology, New Haven, Connecticut
  - Northwestern University Feinberg School Of Medicine, Chicago, Illinois
  - University of Chicago; Hematology/Oncology, Chicago, Illinois
  - University of Iowa Hospital & Clinic; Division of Hematology/Oncology, Iowa City, Iowa
  - Albert B. Chandler Medical Center; University of Kentucky, Lexington, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Chesapeake Urology Research Associates, Towson, Maryland
  - Dana Farber Cancer Inst., Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital., Boston, Massachusetts
  - University Of Michigan, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - MSK @Basking Ridge, Basking Ridge, New Jersey
  - Saint Barnabas Medical Center Cancer Center, Livingston, New Jersey
  - Memorial Sloan-Kettering Cancer Center, Commack, New York
  - Laura and ISAAC Perlmutter Cancer Center at NYU Langone., New York, New York
  - Columbia University Medical Center, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Duke Cancer Center, Durham, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Fairview Hospital; Cleveland Clinic Cancer Center, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Cleveland CL N Coast Cancer Cr, Sandusky, Ohio
  - Abramson Cancer Center; Univ of Pennsylvania, Philadelphia, Pennsylvania
  - Kimmel Cancer Center Thomas Jefferson University, Philadelphia, Pennsylvania
  - Fox Chase-Temple Cancer Center, Philadelphia, Pennsylvania
  - Miriam Hospital, Providence, Rhode Island
  - University of Texas Southwestern, Dallas, Texas
  - Baylor College of Medicine; Gastroenterology, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Virginia, Charlottesville, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington
- Australia (4):
  - Macquarie University Hospital, Macquarie Park, New South Wales
  - Royal Brisbane & Women's Hosp; Cancer Care Serv, Herston, Queensland
  - Monash Medical Centre; Oncology, Clayton, Victoria
  - Austin and Repatriation Medical Centre; Cancer Services, Melbourne, Victoria
- Belgium (4):
  - Institut Jules Bordet, Anderlecht
  - Cliniques Universitaires St-Luc, Brussels
  - UZ Gent, Ghent
  - UZ Leuven Gasthuisberg, Leuven
- Canada (10):
  - Cross Cancer Institute ; Dept of Medical Oncology, Edmonton, Alberta
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - Royal Victoria Hospital, Barrie, Ontario
  - London Regional Cancer Centre, London, Ontario
  - Lakeridge Health Oshawa; Oncology, Oshawa, Ontario
  - The Ottawa Hospital Cancer Centre; Oncology, Ottawa, Ontario
  - North York General Hospital, Toronto, Ontario
  - Sunnybrook Odette Cancer Centre, Toronto, Ontario
  - McGill University; Glen Site; Oncology, Montreal, Quebec
  - CHU de Quebec Hotel-Dieu de Quebec, Québec, Quebec
- China (10):
  - Peking University First Hospital, Beijing
  - Friendship Hospital, Capital Medical University, Beijing
  - Beijing Cancer Hospital, Beijing
  - The Second Affiliated Hospital, Sun Yat-sen University, Guangzhou
  - Jiangsu Province Hospital, Nanjing
  - Jiangsu Cancer Hospital, Nanjing
  - Zhongshan Hospital Fudan University, Shanghai
  - Huashan Hospital Affiliated to Fudan University, Shanghai
  - Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai
- Czechia (4):
  - Masarykuv onkologicky ustav, Brno
  - Fakultni nemocnice Olomouc; Onkologicka klinika, Olomouc
  - Multiscan s.r.o., Pardubice
  - University Hospital Motol; Department of Urology, Prague
- Finland (3):
  - Helsinki University Central Hospital; Urology Clinics, Helsinki
  - Tampere University Hospital; Dept Of Urology, Tampere
  - Turku University Central Hospital; Urology clinic, Turku
- France (14):
  - ICO Paul Papin; Oncologie Medicale., Angers
  - Institut Sainte Catherine;Recherche Clinique, Avignon
  - Hopital Saint Andre, Bordeaux
  - Centre Francois Baclesse; Recherche Clinique, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Leon Berard; Departement Oncologie Medicale, Lyon
  - Centre D'Oncologie de Gentilly; Oncology, Nancy
  - Centre Antoine Lacassagne, Nice
  - Hopital Cochin; Unite Fonctionnelle D Oncologie, Paris
  - Hopital Saint Louis; Oncologie Medicale, Paris
  - Institut Mutualiste Montsouris; Oncologie, Paris
  - Hopital Europeen Georges Pompidou; Service D'Oncologie Medicale, Paris
  - ICO - Site René Gauducheau, Saint-Herblain
  - Institut Claudius Regaud; Departement Oncologie Medicale, Toulouse
- Germany (11):
  - Campus Charitè Mitte Charité Centrum 10. Klinik f.Urologie, Berlin
  - Augusta-Kranken-Anstalt gGmbH; Klinik für Hämatologie, Onkologie & Palliativmedizin, Bochum
  - Universitätsklinikum "Carl Gustav Carus"; Klinik und Poliklinik für Urologie, Dresden
  - Universitätsklinikum Düsseldorf; Urologische Klinik, Düsseldorf
  - Universitätsklinikum der Ruhr-Universität Bochum, Marien-Hospital Herne, Urologische Klinik, Herne
  - Medizinische Fakultät Mannheim, Universitätsklinikum Mannheim, Klinik für Urologie, Mannheim
  - Klinikum rechts der Isar der TU München; Urologische Klinik und Poliklinik, München
  - Universitätsmedizin Rostock, Urologische Klinik und Poliklinik, Rostock
  - Diakonie-Klinikum Stuttgart; Urologische Klinik, Stuttgart
  - Universitätsklinikum Tübingen; Klinik für Urologie, Tübingen
  - Universitätsklinikum Ulm; Klinik für Urologie, Ulm
- Greece (2):
  - Alexandras General Hospital of Athens; Oncology Department, Athens
  - University Hospital of Patras Medical Oncology, Pátrai
- Israel (7):
  - Rambam Health Care Campus; Oncology - Hafia, Hafia
  - Hadassah Ein Karem Hospital; Oncology Dept, Jerusalem
  - Meir Medical Center; Oncology, Kfar Saba
  - Rabin Medical Center; Oncology Dept, Petah Tikva
  - Chaim Sheba Medical Center; Oncology Dept, Ramat Gan
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
  - Assaf Harofeh; Oncology, Ẕerifin
- Italy (10):
  - Az. Osp. Cardarelli; Divisione Di Oncologia, Napoli, Campania
  - ISTITUTO NAZIONALE TUMORI IRCCS FONDAZIONE G. PASCALE; Dipartimento Uro-Ginecologico, Napoli, Campania
  - Azienda Ospedaliero-Universitaria S.Orsola-Malpighi; Unità Operativa Oncologia Medica, Bologna, Emilia-Romagna
  - IRST Istituto Scientifico Romagnolo Per Lo Studio E Cura Dei Tumori, Sede Meldola; Oncologia Medica, Meldola, Emilia-Romagna
  - Azienda Ospedaliera San Camillo Forlanini; Oncologia Medica, Rome, Lazio
  - Irccs Ospedale San Raffaele;Oncologia Medica, Milan, Lombardy
  - Irccs Istituto Europeo Di Oncologia (IEO); Cure Mediche, Milan, Lombardy
  - A.O. UNIVERSITARIA S. LUIGI GONZAGA; Oncologia Medica, Orbassano, Piedmont
  - Azienda USL8 Arezzo-Presidio Ospedaliero 1 San Donato;U.O.C. Oncologia, Arezzo, Tuscany
  - Azienda Ospedaliera S. Maria - Terni; Oncologia, Terni, Umbria
- Japan (17):
  - Nagoya University Hospital; Urology, Aichi
  - Hirosaki University School of Medicine & Hospital; Urology, Aomori
  - Shikoku Cancer Center, Ehime
  - Hiroshima City Hiroshima Citizens Hospital; Urology, Hiroshima
  - National Hospital Organization Hokkaido Cancer Center, Hokkaido
  - University of Tsukuba Hospital, Ibaraki
  - Kyoto University Hospital, Kyoto
  - Iwate Medical University Hospital; Urology, Numakunai
  - Okayama University Hospital, Okayama
  - Osaka University Hospital; Urology, Osaka
  - Kindai University Hospital; Urology, Osaka
  - Saitama Medical University International Medical Center, Saitama
  - Shizuoka Cancer Center; Urology, Shizuoka
  - National Cancer Center Hospital; Urology, Tokyo
  - The University of Tokyo Hospital, Tokyo
  - The Cancer Institute Hospital, JFCR; Urology, Tokyo
  - Kyorin University Hospital, Tokyo
- Netherlands (5):
  - NKI/AvL, Amsterdam
  - VU MEDISCH CENTRUM; Dept. of Medical Oncology, Amsterdam
  - Academ Ziekenhuis Groningen; Medical Oncology, Groningen
  - Erasmus Mc - Daniel Den Hoed Kliniek; Interne Oncologie, Rotterdam
  - St. Antonius locatie Leidsche Rijn, Utrecht
- Poland (5):
  - KO-MED Centra Kliniczne Lublin II, Lublin
  - Szpital Kliniczny im. Heliodora ?wi?cickiego UM w Poznaniu; Oddzia? Chemioterapii, Późna
  - SpecjalistycznySzpital Miejski w Toruniu; Oddzia? Urologii Ogólnej i Onkologicznej, Toru?
  - Szpital Kliniczny Dzieci?tka Jezus; Oddzia? Urologii, Warsaw
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego; Oddzial Urologii i Onkologii, Wroclaw
- Russia (5):
  - SBEI of HPE ?Bashkir State Medical University? of MoH RF, Ufa, Bashkortostan Republic
  - P.A. Herzen Oncological Inst. ; Oncology, Moscow, Moscow Oblast
  - Privolzhsk Regional Medical Center, Nizhny Novgorod, Niznij Novgorod
  - Sverdlovsk Regional Oncology Dispensary; Chemotherapy, Yekaterinburg, Sverdlovsk Oblast
  - Ivanovo Regional Oncology Dispensary, Ivanovo
- Serbia (2):
  - Clinic for Urology; Clinical Hospital Center "Dragisa Misovic-Dedinje", Belgrade
  - Clinical Center of Serbia; Clinic of Urology, Belgrade
- South Korea (3):
  - National Cancer Center, Goyang-si
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (11):
  - Corporacio Sanitaria Parc Tauli; Servicio de Oncologia, Sabadell, Barcelona
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Sant Andreu de la Barca, Barcelona
  - Hospital de Donostia; Servicio de Oncologia Medica, Donostia / San Sebastian, Guipuzcoa
  - Hospital Clinic de Barcelona. Unidad de Nuevas Terapias;Oncology Department, Barcelona
  - Hospital de la Santa Creu i Sant Pau; Servicio de Oncologia, Barcelona
  - Hospital General Universitario Gregorio Marañon; Servicio de Oncologia, Madrid
  - Hospital Ramon y Cajal; Servicio de Oncologia, Madrid
  - Hospital Clinico San Carlos; Servicio de Oncologia, Madrid
  - Hospital Universitario 12 de Octubre; Servicio de Oncologia, Madrid
  - Hospital Universitario La Paz; Servicio de Oncologia, Madrid
  - Instituto Valenciano Oncologia; Oncologia Medica, Valencia
- UniversitätsSpital Zürich; Zentrum für Hämatologie und Onkologie, Klinik für Onkologie, Zurich, Switzerland
- Taiwan (2):
  - Taichung Veterans General Hospital; Division of Urology, Taichung
  - National Taiwan University Hospital, Department of Urology, Taipei
- Turkey (Türkiye) (4):
  - Baskent University Adana Dr. Turgut Noyan Practice and Research Hospital; Medical Oncology, Adana
  - Trakya University Medical Faculty Research And Practice Hospital Medical Oncology Department, Edirne
  - Istanbul Uni Cerrahpasa Medical Faculty Hospital; Medical Oncology, Istanbul
  - Medikal Park Izmir Hospital, Kar??yaka
- Ukraine (3):
  - Regional Clinical Center of Urology and Nephrology n.a. V.I. Shapoval Department of Urology #4, Kharkiv, Kharkiv Governorate
  - CI Dnipropetrovsk CMCH #4 MA of MOHU Ch of Oncology and MR, Dnipropetrovsk
  - GU "Institution of urology of Academy Medical science of Ukraine", Kiev
- United Kingdom (8):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - University Hospitals Bristol NHS Foundation Trust, Bristol
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Barts Health NHS Trust - St Bartholomew's Hospital, London
  - Sarah Cannon Research Institute, London
  - James Cook Uni Hospital, Middlesbrough
  - Royal Preston Hosptial, Preston
  - Southampton General Hospital, Southampton

REFERENCES:
- [Derived] Powles T, Young A, Nimeiri H, Madison RW, Fine A, Zollinger DR, Huang Y, Xu C, Gjoerup OV, Aushev VN, Wu HT, Aleshin A, Carter C, Davarpanah N, Degaonkar V, Gupta P, Mariathasan S, Schleifman E, Assaf ZJ, Oxnard G, Hegde PS. Molecular residual disease detection in resected, muscle-invasive urothelial cancer with a tissue-based comprehensive genomic profiling-informed personalized monitoring assay. Front Oncol. 2023 Jul 31;13:1221718. doi: 10.3389/fonc.2023.1221718. eCollection 2023. PMID 37601688
- [Derived] Bellmunt J, Hussain M, Gschwend JE, Albers P, Oudard S, Castellano D, Daneshmand S, Nishiyama H, Majchrowicz M, Degaonkar V, Shi Y, Mariathasan S, Grivas P, Drakaki A, O'Donnell PH, Rosenberg JE, Geynisman DM, Petrylak DP, Hoffman-Censits J, Bedke J, Kalebasty AR, Zakharia Y, van der Heijden MS, Sternberg CN, Davarpanah NN, Powles T; IMvigor010 Study Group. Adjuvant atezolizumab versus observation in muscle-invasive urothelial carcinoma (IMvigor010): a multicentre, open-label, randomised, phase 3 trial. Lancet Oncol. 2021 Apr;22(4):525-537. doi: 10.1016/S1470-2045(21)00004-8. Epub 2021 Mar 12. PMID 33721560

RESULTS

PARTICIPANT FLOW:
Groups:
- Observation: Participants underwent observation starting on Day 1 for 16 cycles (up to 1 year).
- Atezolizumab: Participants received intravenous (IV) atezolizumab on Day 1 of each 21-day cycle for 16 cycles (up to 1 year).
Period: Overall Study
Arm/Group | Observation | Atezolizumab
Started | 403 | 406
Completed | 171 | 178
Not Completed | 232 | 228
Not completed — Death | 162 | 171
Not completed — Lost to Follow-up | 14 | 12
Not completed — Withdrawal by Subject | 55 | 44
Not completed — Non-specified other | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Observation | Atezolizumab | Total
Number analyzed (Participants) | 403 | 406 | 809
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.9 (9.3) | 66.0 (9.0) | 65.9 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 84 | 171
  Male | 316 | 322 | 638
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 16 | 25
  Not Hispanic or Latino | 357 | 369 | 726
  Unknown or Not Reported | 37 | 21 | 58
Race/Ethnicity, Customized [Number; unit: Number of Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 68 | 64 | 132
  Black or African American | 3 | 3 | 6
  White | 307 | 320 | 627
  Other | 4 | 6 | 10
  Unknown | 21 | 12 | 33

OUTCOME MEASURES:

1. Primary Outcome: Disease-Free Survival (DFS), as Assessed by Investigator
Description: DFS is defined as the time from randomization to the time of first occurrence of a DFS event. DFS events include: local (pelvic) recurrence of UC (including soft tissue and regional lymph nodes); urinary tract recurrence of UC (including all pathological stages and grades); distant metastasis of UC; or death from any cause. Tumor assessment will be performed using radiographic evaluations.
Time Frame: Randomization up to first occurrence of DFS event (up to approximately 50 months)
Population: The ITT population is defined as all randomized patients, whether or not the patient received the assigned treatment (atezolizumab/observation).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Observation | Atezolizumab
Number analyzed (Participants) | 403 | 406
Months | 16.6 [11.2 to 24.8] | 19.4 [15.9 to 24.8]
Statistical Analysis 1: Comparison: Observation vs Atezolizumab; Test type: Superiority; p = 0.2446, Log Rank; Hazard Ratio (HR) = 0.892, 95% CI 2-sided [0.735 to 1.081]

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from randomization to the date of death from any cause, regardless of whether the death occurs during study treatment or following treatment discontinuation.
Time Frame: Randomization until death due to any cause (up to approximately 80 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Observation | Atezolizumab
Number analyzed (Participants) | 403 | 406
Months | 59.0 [47.7 to NA] — Median Overall Survival not reached at the time of final analysis. | 61.4 [47.0 to NA] — Median Overall Survival not reached at the time of final analysis.
Statistical Analysis 1: Comparison: Observation vs Atezolizumab; Stratified analysis based on PDL1 status, tumor stage after resection, and nodal status; Test type: Superiority; p = 0.3172, Log Rank; Hazard Ratio (HR) = 0.897, 95% CI 2-sided [0.726 to 1.109]

3. Secondary Outcome: Disease-Specific Survival (DSS), as Assessed by Investigator
Description: DSS is defined as the time from randomization until the date of death from UC.
Time Frame: Randomization until death due to UC (up to approximately 50 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Observation | Atezolizumab
Number analyzed (Participants) | 403 | 406
Months | NA [NA to NA] — Median has not been reached. | NA [NA to NA] — Median has not been reached.
Statistical Analysis 1: Comparison: Observation vs Atezolizumab; Test type: Superiority — Stratified Analysis; p = 0.2235, Log Rank; Hazard Ratio (HR) = 0.836, 95% CI 2-sided [0.626 to 1.116]

4. Secondary Outcome: Distant Metastasis-Free Survival (DMFS)
Description: DMFS is defined as the time from randomization to the date of diagnosis of distant (that is, non-locoregional) metastases or death from any cause. Tumor assessment will be performed using radiographic evaluations.
Time Frame: Randomization up to diagnosis of distant metastases or death from any cause (up to approximately 50 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Observation | Atezolizumab
Number analyzed (Participants) | 403 | 406
Months | 31.1 [21.7 to 41.4] | 27.5 [22.6 to NA] — Upper bound is not estimable due to insufficient number of subjects with DMFS events.
Statistical Analysis 1: Comparison: Observation vs Atezolizumab; Test type: Superiority — Stratified Analysis; p = 0.4291, Log Rank; Hazard Ratio (HR) = 0.918, 95% CI 2-sided [0.743 to 1.134]

5. Secondary Outcome: Non-Urinary Tract Recurrence-Free Survival (NURFS)
Description: NURFS is defined as the time from randomization to the time of first occurrence of a NURFS event. NURFS events include: local (pelvic) recurrence of UC (including soft tissue and regional lymph nodes); distant metastasis of UC; or death from any cause. Tumor assessment will be performed using radiographic evaluations.
Time Frame: Randomization up to time of first occurrence of a NURFS event (up to approximately 50 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Observation | Atezolizumab
Number analyzed (Participants) | 403 | 406
Months | 19.5 [12.3 to 27.7] | 22.1 [17.2 to 27.6]
Statistical Analysis 1: Comparison: Observation vs Atezolizumab; Test type: Superiority — Stratified Analysis; p = 0.1994, Log Rank; Hazard Ratio (HR) = 0.879, 95% CI 2-sided [0.722 to 1.070]

6. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: Percentage of participants with at least one Adverse Event.
Time Frame: Screening up to approximately 80 months
Population: The safety population is defined as patients who received at least one dose of atezolizumab, and all patients who did not receive any dose of atezolizumab who had at least one post-baseline safety assessment (e.g.,adverse event, lab, vital signs, ECG, etc.), regardless of their assigned treatment (atezolizumab/observation).
Measure: Number; unit: Percentage of Participants
Arm/Group | Observation | Atezolizumab
Number analyzed (Participants) | 398 | 390
Percentage of Participants | 79.1 | 94.4

7. Secondary Outcome: Percentage of Participants With Anti-Therapeutic Antibodies (ATAs) to Atezolizumab
Description: Percentage of participants with anti-therapeutic antibodies to atezolizumab.
Time Frame: Baseline up to approximately 50 months
Population: The anti-drug antibodies (ADA)-evaluable population is defined as all patients treated with atezolizumab who have at least one post-baseline ADA result.
Measure: Number; unit: Percentage of Participants
Arm/Group | Atezolizumab
Number analyzed (Participants) | 375
Percentage of Participants | 29.3

8. Secondary Outcome: EuroQol 5-Dimension 5-Level (EQ-5D-5L) Visual Analogue Scale Score
Description: The EQ-5D-5L is a generic preference-based HRQoL questionnaire that provides a single index value for health status and is used to inform pharmacoeconomic evaluations and to measure general health status. Visual analog scale (VAS) allows the patient to indicate, on a scale of 0-100, how his or her health is on the day of assessment, with 100 being the "best imaginable health state" and 0 being the "worst imaginable health state."
Time Frame: Day 1 of Cycle 1 up to approximately 50 months (Cycle length = 21 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Observation | Atezolizumab
Number analyzed (Participants) | 403 | 406
Score on scale
  Cycle 1 Day 1: number analyzed (Participants) | 375 | 375
  Cycle 1 Day 1 | 77.41 (15.74) | 78.89 (16.13)
  Cycle 3 Day 1: number analyzed (Participants) | 349 | 338
  Cycle 3 Day 1 | 78.64 (15.73) | 81.05 (14.96)
  Cycle 5 Day 1: number analyzed (Participants) | 277 | 295
  Cycle 5 Day 1 | 79.94 (16.32) | 81.95 (14.32)
  Cycle 7 Day 1: number analyzed (Participants) | 259 | 267
  Cycle 7 Day 1 | 80.81 (16.37) | 82.39 (14.43)
  Cycle 9 Day 1: number analyzed (Participants) | 228 | 250
  Cycle 9 Day 1 | 81.24 (15.70) | 82.06 (15.34)
  Cycle 11 Day 1: number analyzed (Participants) | 209 | 220
  Cycle 11 Day 1 | 81.39 (17.02) | 82.81 (14.96)
  Cycle 13 Day 1: number analyzed (Participants) | 190 | 216
  Cycle 13 Day 1 | 81.39 (16.99) | 82.59 (14.81)
  Cycle 15 Day 1: number analyzed (Participants) | 187 | 180
  Cycle 15 Day 1 | 82.78 (16.01) | 83.67 (14.47)
  Treatment Discontinuation: number analyzed (Participants) | 176 | 219
  Treatment Discontinuation | 82.68 (16.19) | 81.91 (15.96)

9. Secondary Outcome: Minimum Observed Serum Atezolizumab Concentration (Cmin)
Description: Minimum observed serum atezolizumab concentration (Cmin) prior to infusion on Day 1 of Cycles 1, 2, 3, and 4; every 8 cycles starting on Cycle 8; at treatment discontinuation; and at 120 days after the last dose of atezolizumab.
Time Frame: Pre-dose (Hour 0) on Day 1 of Cycles 1, 2, 3, 4, every 8 cycles from Cycle 8, at treatment discontinuation, 120 days after treatment discontinuation (up to approximately 50 months))(Cycle length = 21 days)
Population: The pharmacokinetic-evaluable population is defined as all patients who received any dose of atezolizumab and who have evaluable pharmacokinetic (PK) samples.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Atezolizumab
Number analyzed (Participants) | 380
µg/mL
  Cycle 2 Day 1: number analyzed (Participants) | 355
  Cycle 2 Day 1 | 78.4 (25.2)
  Cycle 3 Day 1: number analyzed (Participants) | 335
  Cycle 3 Day 1 | 125 (46.0)
  Cycle 4 Day 1: number analyzed (Participants) | 323
  Cycle 4 Day 1 | 152 (71.1)
  Cycle 8 Day 1: number analyzed (Participants) | 254
  Cycle 8 Day 1 | 203 (92.0)
  Cycle 16 Day 1: number analyzed (Participants) | 163
  Cycle 16 Day 1 | 225 (106)
  Day 120 Post Last Dose MPDL3280A: number analyzed (Participants) | 195
  Day 120 Post Last Dose MPDL3280A | 15.9 (19.5)
  Study Drug or Study Phase Comp or Early Disc: number analyzed (Participants) | 277
  Study Drug or Study Phase Comp or Early Disc | 164 (106)

10. Secondary Outcome: Maximum Observed Serum Atezolizumab Concentration (Cmax)
Description: Maximum observed serum atezolizumab concentration (Cmax) after infusion on Day 1 of Cycle 1.
Time Frame: Day 1 of Cycle 1 (Cycle length = 21 days)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Atezolizumab
Number analyzed (Participants) | 300
µg/mL | 365 (121)

ADVERSE EVENTS:
Time Frame: From the first study drug to the data cutoff date: 14 June 2022 (up to 80 months)
Description: Safety-evaluable population for atezolizumab included patients who received at least 1 dose of atezolizumab. Safety-evaluable population for observation included patients randomized to observation who had at least 1 post-baseline safety assessment. All-cause mortality reported for deaths that occurred during study based on ITT, which included all randomized patients.
Arm/Group | OBSERVATION | ATEZOLIZUMAB
All-Cause Mortality (participants affected / at risk) | 162/403 | 171/406
Serious Adverse Events (participants affected / at risk) | 72/398 | 122/390
Other Adverse Events (participants affected / at risk) | 234/398 | 324/390
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OBSERVATION (N=398) | ATEZOLIZUMAB (N=390)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Hypophysitis (Endocrine disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 4 (4)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 5 (5)
Enterovesical fistula (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hernial eventration (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 1 (1)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 4 (5)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Mechanical ileus (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 1 (1)
Small intestine ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 3 (3)
Hernia pain (General disorders) | 1 (1) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Lithiasis (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 3 (3) | 11 (11)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 2 (3)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic haematoma (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 2 (2)
Systemic immune activation (Immune system disorders) | 0 (0) | 2 (2)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Bacterial sepsis (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Diabetic foot infection (Infections and infestations) | 0 (0) | 1 (1)
Escherichia sepsis (Infections and infestations) | 1 (1) | 0 (0)
Febrile infection (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 1 (1)
Kidney infection (Infections and infestations) | 1 (1) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Neuroborreliosis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 4 (4)
Pyelonephritis (Infections and infestations) | 9 (11) | 12 (16)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 1 (2)
Pyelonephritis chronic (Infections and infestations) | 0 (0) | 1 (1)
Renal abscess (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 3 (5)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 19 (21) | 30 (41)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 1 (1)
Urosepsis (Infections and infestations) | 3 (3) | 1 (1)
Vascular device infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Incision site impaired healing (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Stoma obstruction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Stomal hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ureteric anastomosis complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Urostomy complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Device dislocation (Product Issues) | 1 (1) | 0 (0)
Device occlusion (Product Issues) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 8 (8)
Autoimmune nephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 1 (1)
Nephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (3)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 1 (2) | 1 (1)
Ureteric stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 2 (2)
Urinoma (Renal and urinary disorders) | 1 (1) | 0 (0)
Vesicoureteric reflux (Renal and urinary disorders) | 0 (0) | 1 (1)
Female genital tract fistula (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Lymphocele (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Immune-mediated neurological disorder (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OBSERVATION (N=398) | ATEZOLIZUMAB (N=390)
Anaemia (Blood and lymphatic system disorders) | 32 (34) | 42 (53)
Hypothyroidism (Endocrine disorders) | 0 (0) | 35 (38)
Abdominal pain (Gastrointestinal disorders) | 29 (32) | 31 (39)
Constipation (Gastrointestinal disorders) | 39 (40) | 51 (60)
Diarrhoea (Gastrointestinal disorders) | 25 (29) | 81 (104)
Nausea (Gastrointestinal disorders) | 20 (21) | 52 (60)
Vomiting (Gastrointestinal disorders) | 14 (16) | 26 (34)
Asthenia (General disorders) | 16 (16) | 35 (41)
Chills (General disorders) | 7 (9) | 23 (25)
Fatigue (General disorders) | 43 (50) | 89 (118)
Oedema peripheral (General disorders) | 23 (26) | 34 (39)
Pyrexia (General disorders) | 30 (43) | 71 (90)
Upper respiratory tract infection (Infections and infestations) | 18 (19) | 21 (27)
Urinary tract infection (Infections and infestations) | 59 (84) | 63 (88)
Alanine aminotransferase increased (Investigations) | 7 (8) | 24 (32)
Aspartate aminotransferase increased (Investigations) | 5 (6) | 20 (25)
Blood alkaline phosphatase increased (Investigations) | 8 (8) | 20 (29)
Blood creatinine increased (Investigations) | 17 (20) | 37 (42)
Decreased appetite (Metabolism and nutrition disorders) | 20 (21) | 45 (54)
Arthralgia (Musculoskeletal and connective tissue disorders) | 26 (29) | 53 (62)
Back pain (Musculoskeletal and connective tissue disorders) | 44 (51) | 26 (30)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (8) | 21 (30)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (9) | 22 (29)
Dizziness (Nervous system disorders) | 11 (11) | 20 (22)
Headache (Nervous system disorders) | 8 (8) | 35 (39)
Cough (Respiratory, thoracic and mediastinal disorders) | 23 (23) | 47 (60)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 27 (33)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 29 (30)
Pruritus (Skin and subcutaneous tissue disorders) | 10 (15) | 92 (113)
Rash (Skin and subcutaneous tissue disorders) | 5 (6) | 38 (48)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-04-13): https://cdn.clinicaltrials.gov/large-docs/31/NCT02450331/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/31/NCT02450331/SAP_001.pdf